CLINICAL TRIAL: NCT03907644
Title: Frontoparietal Synchronization to Modulate Drug Craving in Opioid Use Disorder: A Randomized Experimental Trial
Brief Title: Frontoparietal Synchronization to Modulate Drug Craving in Opioid Use Disorder
Acronym: FPS_Opioid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019-001-00
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active FPS (Experimental): We use Starstim AC (alternative current) -Stimulator R32. FPS protocol will be used with 20 minutes 2mAmp 6 Hz tACS to the middle frontal gyrus (DLPFC, F4 in EEG electrodes with 10-20 system measurement) and inferior parietal cortex (IPC, P4), as the main nodes of the frontoparietal network, in synchronous oscillation. The 4 return electrodes will receive 0.5 mAmp each around each active electrode (High Definition Montage). The electrodes are silver/silver chloride that are wet with conductive gel. We will use surface landmarks and EEG caps on the head to place the electrodes, which are held in place by head caps with holes indicating places for electrode positioning.
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)
- Sham FPS (Sham Comparator): In the sham stimulation mode, the device shows pseudorandom numbers on the screen that look like real stimulation is being delivered. The device gives a low level of stimulation at the very beginning and at the very end of the stimulation session (30 seconds ramp up and 30 seconds ramp down) in order to recreate the feeling of tingling that subjects perceive at the beginning and end of real stimulation.
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation (tACS) — The tACS stimulator delivers very low (2mAmp) current with surface electrodes to the skull.

SUMMARY:
Opioid use disorder (OUD) is among the costliest and deadliest substance use disorders (SUDs) in the US and world-wide. Opioids were involved in 42,249 deaths in the US in 2016, which were more than deaths due to road accidents and gun violence combined. Opioid overdose deaths were five times higher in 2016 than 1999. Meanwhile, the treatment options for OUD are limited and long-term efficacy is poor. There is a hope that recent advances in understanding of the cognitive neuroscience underlying addictive behavior, like drug craving and its regulatory processes, can bring new opportunities for more effective and personalized treatment options for OUD. Drug craving is the signature aspect of OUD as well as other SUDs which has been associated with continued drug use and relapse. In previous studies, the investigators have shown significant response to drug related cues in both frontoparietal and limbic areas including amygdala and ventral striatum. In a recent pilot study, the investigators showed significant lower connectivity between amygdala and frontoparietal areas, including dorsolateral prefrontal cortex (DLPFC) and inferior parietal cortex (IPC), major nodes of the executive control network (ECN), in patients with OUD compared with healthy controls. The central role of the ECN is to perform top down regulation of subcortical limbic areas during self-control, emotion-regulation, and response- inhibition tasks. These processes are well known to be affected in different psychopathologies including SUDs. There is a growing body of evidence that external frontoparietal synchronization (FPS) with transcranial alternating current stimulation (tACS) can potentially modulate connectivity within ECN and between ECN and limbic areas. This may improve some aspects of executive function and top down regulation. tACS is a low-cost and scalable non-invasive brain stimulation technology without any serious side effects. The procedure involves the transcranial delivery of low levels of alternating current (0.1-2 mAmp) in different frequencies through the skull into the brain with both online and long-term offline effects. This trial is the first combined tACS/fMRI study to examine the acute offline effects of FPS on neural substrates underlying drug induced craving. We hypothesize that FPS amplifies the ECN top-down modulatory role via its connectivity to other cortical-subcortical areas. In this experimental design, the investigators will recruit 60 people with OUD during the early abstinence phase in a residential setting divided into two parallel arms with active and sham FPS tACS. Each subject will undergo resting state and task based (drug cue exposure paradigm) functional MRI pre and post FPS. The investigators will also conduct individual difference analyses to explore the potential predictors for FPS response, including pre-FPS top-down connectivity measures of ECN and other subjective, clinical, behavioral, structural, and functional variables. The results of this study will provide mechanistic neuroscience-based evidence for the efficacy of FPS and will advance the field towards precision addiction medicine.

DETAILED DESCRIPTION:
A. Background:

Opioid use disorder (OUD) is among the costliest and deadliest substance use disorders (SUDs) in the US and world-wide. Opioids (including prescription opioids, heroin, and fentanyl) were involved in more than 42,000 deaths in 2016 in US, more than any year on record and accounting for more deaths than due to road accidents and gun violence combined1. Over 4.3 million Americans engaged in non-medical use of prescription opioids each month and 4.8 million people have used heroin at some point in their lives. From each year since 2002, past month heroin use, past year heroin use, and heroin use disorder have increased among 18-25 years old. Among new heroin users, approximately three out of four reported using prescription opioids prior to using heroin. Available treatment options for OUD are limited and long-term efficacy to return to a normal life is very low. During the last two decades, advancements in human neuroscience research have provided new hope for targeting neurocognitive processes underlying drug addictions, including OUD, to introduce new therapeutic interventions. In reality, however, neuroscience has played a very minimal role, if any, in changing clinical practices for OUD, until now.

Although DSM V has added "drug craving" as a criterion for SUDs, it has been well-known as a core process in drug dependence and addiction for many years. Exposure to drug-related cues to induce drug craving, which is called "Cue Induced Craving" or "CIC", is one of the main paradigms used to study the drug craving phenomenon2. There are many studies that have shown CIC to be a valid core construct for continued drug use and relapse. Therefore, reduction of CIC is now one of the main targets for enhancing substance use recovery2. Different brain areas and networks are involved in CIC. In particular, top down modulation by frontoparietal areas involved in the executive control network (ECN) including dorsolateral prefrontal cortex (DLPFC), and inferior parietal cortex (IPC), over subcortical areas such as ventral striatum (VSt) and amygdala, is thought to be the critical process underlying CIC. Failure of top down modulation by ECN in relation to other large-scale networks is reported to be a predictor of relapse among both cocaine and heroin users. Furthermore, improvement in ECN top-down regulation has been reported in trials with medications that reduce drug craving3. This is in line with current evidence from animal models for the central role of frontoparietal network in top-down attention and executive control. It is frequently reported that coherence in the theta band (4-8 Hz) within the frontoparietal network plays a central role in executive functions including working memory and cognitive control. There is a growing body of evidence that transcranial alternating current stimulation (tACS) can increase this coherence, entrain ECN connectivity and improve its function. tACS is a device-based technology employed to change cortical oscillations by applying a very weak (0.1 to 2mAmp) alternating current over the skull. In vivo studies show that tACS can modulate ongoing neural rhythms by shifting spike timing and firing rates towards the stimulation frequency (external synchronization)4. Meanwhile, it is strongly proposed that synchronized oscillation plays the major role in communication and connection between nodes within a network5. Based on this background, there is hope that multisite tACS (mtACS), with synchronized current delivered to the sites (network nodes), can offer the potential to enhance connectivity between nodes of these large-scale networks. FrontoParietal Synchronization (FPS), defined as a double site, DLPFC and IPC, tACS both with in-phase (synchronic) oscillatory electric current, more frequently in the theta or alpha bands, has received particular attention among other mtACS methods. The goal of FPS is to improve ECN connectivity and improve functions like working memory6-8 and attention control9. Most tACS studies have explored the online effects of synchronization. However, recent evidence for the long-lasting entraining effect of tACS after termination of stimulation (offline effect) has increased the potential for meaningful clinical applications. Nevertheless, there are no published fMRI studies to date (Dec 2018) that have aimed to delineate how FPS might modulate top-down ECN regulatory control over the amygdala and ventral striatum. The overall aim of the proposed research is thus to determine whether FPS can amplify top down modulation of ECN over subcortical-limbic areas (VSt and Amygdala) during CIC among people with OUD. Furthermore, the investigators will explore whether connectivity between these areas before FPS along with other clinical and behavioral factors can predict inter- individual differences in subjective response to FPS in CIC. This line of research will provide a mechanistic background to use context-dependent tACS to enhance cognitive control in drug craving to improve long term drug addiction treatment outcomes.

B. Significance:

This study combines an active intervention with behavioral and neuroimaging assessments in people suffering from OUD, a target population in the US with extensive need for new treatment options. tACS involves simple and low-cost technology without any significant side effects that is largely scalable as a potential non-invasive therapeutic tool to help people during addiction recovery. Results will help provide a mechanism for how transcranial electrical current interventions can affect neurocognitive processes involved in drug addiction with the long-term goal of improving treatment outcomes.

C. Innovation:

For the first time, the investigators will be able to delineate the mechanistic neural substrates that are important for the efficacy of FPS for OUD using both task-based and resting state functional neuroimaging methods. Moreover, using an individual differences approach, the investigators will be able to identify prognostic biomarkers for the efficacy of FPS among individuals with OUD, advancing the field towards precision addiction medicine.

D. Specific Aims:

1. To determine whether FPS changes ECN (DLPFC, and IPC) and limbic (VSt and Amygdala) task (CIC) and resting state connectivity (neural response to FPS) in OUD
2. To determine whether FPS changes subjective self-report of craving (subjective response to FPS)
3. To explore whether pre-FPS ECN-limbic connectivity predicts neural and/or subjective response to FPS
4. To explore which of (a) subjective, (b) clinical, (c) behavioral, (d) structural, or (e) neural circuits measures predict neural and/or subjective response to FPS

E. Research Design and Methods:

This is an experimental study of a single session FPS in medically healthy male individuals with opioid use disorder (OUD). Subjects will be screened and enrolled from residential abstinence-based treatment centers (like 12&12 Addiction Treatment Center) or inpatient programs (like Laureate Psychiatric Clinic and Hospital). Effects of FPS on drug craving will be assessed by both questionnaires and resting state and task-based fMRI.

Screening: The substance use core protocol (LIBR protocol #2018-012, PI: Martin Paulus), which includes multi-level baseline assessment will be used to screen potential subjects at addiction treatment programs in Tulsa (i.e., 12 & 12, LPCH and etc.). Participants who complete that protocol and meet criteria for the current study will be invited to participate. 12 & 12 is a leader in the substance abuse and addiction treatment and recovery fields and the largest non-profit addiction treatment facility in a four-state area offering residential and outpatient treatment services for both substance abuse and co-occurring conditions (those with a mental health issue as well as an addiction diagnosis). It is located less than 4 miles from Laureate Institute for Brain Research. Laureate Psychiatric Clinic and Hospital (LPCH) is basically attached to LIBR and offer both inpatient and outpatient treatment services for drug addiction. All potential subjects will be introduced by the clinical team at the treatment programs and then be screened by the trained study staff or the PI to determine whether they meet any exclusion criteria such as any major medical or psychiatric illness that would preclude the use of tACS and or fMRI. Subjects will be screened for psychiatric disorders by the trained staff with Mini International Neuropsychiatric Interview.

Consent: The purpose, content, duration, and expected risks and benefits of the study will be reviewed with each potential subject by the trained study staff. If they pass the screening interview, written consent will also be obtained before subjects can participate in any portion of the study. The actual consent form will either be given to the potential participant by mail, email or in-person, depending on their preference. Subjects will be encouraged to be open with the investigator and/or staff about any questions or concerns they have either before, during, or after the study.

Enrollment: Sixty subjects with OUD will be recruited from residential or inpatient addiction treatment programs in Tulsa in their first weeks of abstinence after being medically stabilized. Participants will undergo screening and baseline assessments using self-report and clinical assessments. Eligible participants will be allocated to either active or sham stimulation arms in. Participants in the active arm will receive 20 minutes FPS on right ECN. The right ECN is selected as its contribution is dominant among people with SUD 10. Moreover, right FPS has been reported to have more pronounced effects on executive functions. Resting state (rs) and task-based fMRI (pictorial opioid cue exposure, block-designed) and EEG (electroencephalography) will be done immediately before and after active or sham FPS. Drug craving will be assessed with a single item 0-100 VAS (visual analogue scale) question at multiple time points before and after imaging and FPS. Subjective and neural response to drug cue exposure in prefrontal cortical areas and subcortical-limbic areas (craving>neutral activations) and their connectivity during resting state will be assessed before and after FPS with contrasts made between active and sham stimulation with a random effects model.

F. Hypotheses and Statistical Methods The basic image processing will be done with the AFNI software package. Subject-level analyses on rs- and task-based fMRI data will generate functional connectivity z-scores and beta maps, respectively for group-level analyses.

For the primary outcome measure and first secondary outcome measure, subjective report and neural response to drug cue exposure in prefrontal cortical areas and subcortical-limbic areas (Fig 1) and their connectivity during resting state will be assessed before and after FPS with contrasts made between active and sham stimulation with random effect. Beta maps will be used to evaluate drug-cue reactivity at regions of interest (ROIs) by mixed-effects models (AFNI 3dMEMA); multiple comparisons will be corrected by false-discovery rate (FDR) or cluster level thresholds (AFNI 3dClustSim). The investigators hypothesize that FPS significantly reduces subjective reports of craving, increase activations in the prefrontal cortical areas and insula, decreases activations in the ventral striatum and amygdala and increase top-down connectivity between cortical and subcortical areas within ROIs.

For the other secondary outcome measures, the investigators will use a linear regression model to identify factors contributing to response to FPS in the active arm. The investigators hypothesize that higher baseline top-down connectivity will have a significant effect on the higher FPS effects in reducing activations in the subcortical areas. The investigators also hypothesize that higher current intensity in the cortical areas would have significant positive effects on the both subjective and neural responses to the FPS.

For the exploratory outcome measures, an exploratory regularized regression model (elastic net) will be employed to define major prognostic factors for response to FPS in the active arm of the study. This model will be validated with one-leave-out cross validation within this dataset and will be validated with subsequent test datasets in the future studies.

The proposed sample size of 30 participants per arm will provide 80% power to detect an effect size (Cohen's d) of 0.74 for changes in drug-cue reactivity between arms at a two-sided 0.05 significance level in a two-sample t-test.

G. Gender/Minority/Pediatric Inclusion for Research The investigators will include male participants age 18 and older. Women will not be included in this preliminary study to control for the effects of hormonal changes on brain plasticity induced by FPS. Subjects will be recruited without any predilection for any racial or ethnic groups.

H. Subject Risks

Assessments: Risks and general protections against risk: The main risk to the subjects is that assessments with self-reports, interviews and cognitive tasks take time. The assessments being used in this study are the same as those used in different studies at Laureate Institute for Brain Research. Some people may find some of the questions to be too personal but the subjects always have the option of not answering any questions.

FPS: Risks and general protections against risk: Subjects will be fully informed about the foreseeable risks and discomforts associated with participation in this study.

1. Headaches/itching/paresthesia. Headaches, itching, and paresthesia are generally very mild with FPS and are limited to the actual treatment duration. Since skin nerves habituate to the electrical stimulation rather quickly, most subjects are not aware of the stimulation after about the first 1-minute. This is what allows sham stimulation to be effectively masked. More persistent headache can be treated with acetaminophen or ibuprofen. The range of stimulation intensities for human studies of FPS is usually 1-2mAmps as the investigators do in this study.
2. Skin irritation. Skin redness is common with FPS studies because the electrical stimulation increases local blood flow under the electrodes. This redness should dissipate within 30-minutes or less. There should be no evidence of redness or skin breakdown before the FPS application.

The consent forms describe these risks and discomforts clearly. Patients must know that they have the option to withdraw from the study at any time. Withdrawal from this study can be done without consequence. The investigators may also choose to terminate a participant from this study, if they suffer a severe adverse event, do not follow study requirements, or feel that continued participation would put the person at a greater risk than indicated.

Drug Cue Exposure: Risks and general protections against risk: Drug cue exposure is a conventional method in experimental addiction studies. Functional neuroimaging with MRI (fMRI) with drug cue exposure tasks is a routine method to activate and depict neurocircuits involved in drug craving. There are over 300 published studies indexed at the National Library of Medicine's website (www.pubmed.com) with drug cue exposure fMRI among drug users. The only risk that is associated with these paradigms other than minimal risks associated with fMRI in general is the increased level of drug craving among participants. In this study, like other studies in the field, the investigators will assess the level of craving after the cue exposure sessions inside or outside MRI scanner to ensure that subjects will not leave the center with a significant level of craving. Different craving reduction methods, such as relaxation, distraction or reappraisal will be instructed to the study staff to help participants to calm down any potential craving. After assurance that the participants are in stable condition, they will be escorted back to the treatment program or other facilities with minimum risk for access to drugs.

I. Benefits versus Risk In accordance to the principle of beneficence, research should maintain a favorable balance of benefit to risk. The proposed FPS parameters in OUD patients in this protocol fall within a Class II classification of benefit-risk ratio. That is, FPS, as used here, is of potential, but unproven benefit. Given the investigators experience, the FDA approval of a tDCS (transcranial direct current stimulation) /tACS (transcranial alternating current stimulation) device that is actively marketed to the public, and experience of other tDCS/tACS laboratories, to date, the tDCS/tACS parameters used in this protocol are safe and constitute a 'minimal risk' application.

J. Data and Safety Monitoring Plan The risk for adverse events is minimal. No medication, therapeutic decision or investigational device is made based on the results of these studies. Participants may experience some discomfort upon discussing their symptoms with staff and receiving unanticipated information about diagnosis. Participants may find it difficult to participate in detailed ratings. Any unanticipated adverse events will be reported immediately to the IRB of record and Laureate Institute for Brain Research Human Protection Administrator at (918) 502-5155 or via email at hpa@laureateinstitute.org.

Each subject is given a unique identifier with a code. Information for each participant is entered into the Laureate Institute for Brain Research subject database and they are automatically given a LIBR number. The code key that links the unique identifier to the subjects' names is kept in a separate file. All data analysis is performed on de-identified data. Other than the principal investigators, there is no need for personally identifying information to be known to other investigators.

The electronic data will be kept in a firewalled and password protected database on a secure server managed by LIBR. Vanderbilt University, with collaboration from a consortium of institutional partners, has developed a software toolset and workflow methodology for electronic collection and management of research and clinical trial data. REDCap (Research Electronic Data Capture) data collection projects rely on a thorough study-specific data dictionary defined in an iterative self-documenting process by all members of the research team with planning assistance from the information technology staff. The iterative development and testing process results in a well-planned data collection strategy for individual studies. REDCap servers are housed in a local data center at Laureate Institute for Brain Research and all web-based information transmission is encrypted. REDCap was developed specifically around HIPAA-Security guidelines and is recommended to LIBR researchers by both the investigators' Privacy Office and the Western Institutional Review Board (WIRB). REDCap has been disseminated for use locally at other institutions and currently supports 240+ academic/non-profit consortium partners on six continents and over 26,000 research end-users (www.project-redcap.org).

Subjects will not be identified in any reports or publications. If the PI leaves LIBR, and agreement will be made between LIBR and the PI new institution to transfer the data so that the study can continue.

Study information will be made available to the subjects when there has been sufficient data analysis to make reasonable aggregate conclusions. The investigators can share general study characteristics (how many people were recruited, age, primary disorder etc.) early in the process but the investigators do not share study results with subjects until the quality of the data is close to publication level.

K. CONFIDENTIALITY Records of the participant's participation in this study will be held confidential except as disclosure is required by law or as described in the informed consent document (under "Confidentiality"). The researchers will make every effort to minimize the risk of breach of confidentiality and a Certificate of Confidentiality will be obtained from NIH to further protect the subject. The study doctor, the sponsor or persons working on behalf of the sponsor, and under certain circumstances, the United States Food and Drug Administration (FDA) and WIRB will be able to inspect and copy confidential study-related records that identify the subject by name. Therefore, absolute confidentiality cannot be guaranteed. If the results of this study are published or presented at meetings, the subject will not be identified. Paper copies of consents, screening forms, the Research Privacy Form, and any other forms, testing results or papers containing Personally Identifiable Information (PII) will be stored in a secured medical records room or electronically with access granted only to authorized personnel.

The study PIs, the sponsor or persons working on behalf of the sponsor, and under certain circumstances, the United States Food and Drug Administration (FDA) and the Institutional Review Board (IRB) will be able to inspect and copy confidential study-related records which identify the subject by name. Therefore, absolute confidentiality cannot be guaranteed. If the results of this study are published or presented at meetings, the subject will not be identified.

Electronic copies of consents, screening forms, and any other forms, testing results or papers containing Personally Identifiable Information (PII) will be stored on a password protected electronic database with access granted only to authorized personnel.

ELIGIBILITY:
Inclusion criteria:

1. Male
2. Age ≥18 and <61 years old
3. English speaking
4. Diagnosed with Opioid Use Disorder (last 12 months) based on the structured interview (DSM V)
5. Being abstinent from opioid in an addiction treatment program for at least 3 days based on medical records or self-report
6. Positive response to Opioid cue-reactivity screening (OCS)
7. Willing and capable of interacting with the informed consent process

Exclusion criteria:

1. Unwillingness or inability to complete any of the major aspects of the study protocol, including magnetic resonance imaging (i.e., due to claustrophobia), drug cue rating, or behavioral assessment.
2. Abstinence from opioid for more than 6 months based on self-report
3. Schizophrenia or bipolar disorder based on the MINI interview
4. Active suicidal ideation with intent or plan determined by self-report or assessment by PI or study staff during the initial screening or any other phase of the study
5. Positive drug test for amphetamines, opioids, cannabis, alcohol, phencyclidine, or cocaine confirmed by breath analyzer and urine tests
6. Any active skin disorder that affects skin integrity of the scalp
7. Having any condition that would preclude undergoing an fMRI scan or FPS (tACS) stimulation based on the fMRI safety and transcranial electrical stimulation safety checklists
8. Unstable medical disorder reported in subject's medical history or by a clinician assessment
9. History of seizure
10. Non-correctable vision or hearing problems.
11. Any other condition the PI or study staff feel would put the subject at risk for entering the study

Ages: 18 Years to 61 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Drug Cue Reactivity BOLD Signal in fMRI from before to after Intervention | Immediate before and immediate after intervention
  Drug Cue Reactivity BOLD Signal is measured as average blood oxygen level dependent (BOLD) signal difference with voxel-wise analysis in the regions of interests (ROIs) (prefrontal cortex parcels, insula segments, striatum nuclei, thalamus nuclei and extended amygdala nuclei) in craving > neutral contrast in drug cue exposure fMRI task with blocks of neutral and drug related images

SECONDARY OUTCOMES:
Change in Drug Cue Reactivity Self-Report from before to after Intervention | Immediate before and immediate after intervention
  Drug cue reactivity self-report is measured as the difference in subjective response to "On a scale of 0-100, How much drug craving are you experiencing right now" measured on a visual analog scale (0-100) before and after drug cue exposure fMRI task. Higher reduction in this outcome in active group compared to sham means a better outcome.
Change in Cortical-Subcortical Connectivity in Resting State fMRI from before to after Intervention | Immediate before and immediate after intervention
  Cortical-Subcortical Connectivity is measured as correlation between resting-state average blood oxygen level dependent (BOLD) signal time series in subcortical ROIs and voxels within prefrontal cortex and Insula

OTHER OUTCOMES:
Change in Cortical-Subcortical Task-based Connectivity in Cue Exposure fMRI from before to after Intervention | Immediate before and immediate after intervention
  Cortical-subcortical task-based connectivity in cue exposure fMRI is measured as psychophysiological interaction (PPI) between average blood oxygen level dependent (BOLD) signal time series in subcortical ROIs and voxels within prefrontal cortex and insula, using craving > neutral contrast regressor
Change in RAI in Resting State fMRI from before to after Intervention | Immediate before and immediate after intervention
  Resource Allocation Index (RAI) is measured with the correlation among default mode network (DMN), saliency network (SN) and Executive Control Network (ECN) in resting state fMRI based on Lerman, et al., 2014.
Change in Area Under Electrode Connectivity in Resting State fMRI from before to after Intervention | Immediate before and immediate after intervention
  Area under electrode connectivity is measured with voxel-wise correlation between average blood oxygen level dependent (BOLD) signal in the cortical area under the Anode and Cathode electrodes and whole brain
Change in Area Under Electrode Task-based Connectivity in Cue Exposure fMRI from before to after Intervention | Immediate before and immediate after intervention
  Area under electrode task-based connectivity is measured with voxel-wise Psychophysiological Interaction (PPI) between average blood oxygen level dependent (BOLD) signal in the cortical area under the Anode and Cathode electrodes and whole brain using craving > neutral contrast regressor in block-design drug cue exposure fMRI task
Change in Momentary Craving Self-Report from before to after Intervention | Immediate before and immediate after intervention
  Momentary craving self-report is assessed with subjective response to "On a scale of 0-100, How much drug craving are you experiencing right now" measured on a visual analog scale (0-100)
Change in Drug Cue Control Response from before to after Intervention | Immediate before and immediate after intervention
  Drug cue control response is measured as the difference in subjective response to "On a scale of 0-100, How much CONTROL over your drug craving are you experiencing right now" measured on a visual analog scale (0-100) before and after drug cue exposure fMRI task

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No